CLINICAL TRIAL: NCT02794220
Title: A Randomised, 4-way Crossover, Relative Bioavailability Study of Nicotine Delivered by an Electronic Cigarette, Nicorette® Inhalator and Cigarette Smoking
Brief Title: A Study of Blood Levels of Nicotine Following an Electronic Cigarette
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Simbec Research (Industry)
Collaborators: CN creative (Unknown)
Responsible Party: Principal Investigator, Girish Sharma, MBBS, Simbec Research
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: RD 655/25310
Record Dates: First submitted 2016-06-03; First posted 2016-06-09 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-06

CONDITIONS: Nicotine Replacement Therapy
Keywords: E-cigarette; healthy volunteer study; Pharmacokinetics; Nicorette
MeSH Terms: conditions — Vaping | interventions — Tobacco Products

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- CN Electronic cigarette 10 mg (Experimental): 10 mg strength
  - Administration once every hour for a total of 4 hours.
  Interventions: Device: CN electronic cigarette 10 mg
- CN Electronic cigarette 15 mg (Experimental): 15 mg strength
  - Administration once every hour for a total of 4 hours.
  Interventions: Device: CN electronic cigarette 15 mg
- Nicorette Inhalator 15 mg (Active Comparator): 15 mg strength
  - Administration once every hour for a total of 4 hours.
  Interventions: Device: Nicorette Inhalator 15 mg
- Cigarette (Active Comparator): Subjects will all smoke the same brand.
  - Administration once every hour for a total of 4 hours.
  Interventions: Other: Cigarette

INTERVENTIONS:
Device: CN electronic cigarette 10 mg — Inhalation
  Arms: CN Electronic cigarette 10 mg
Device: CN electronic cigarette 15 mg — Inhalation
  Arms: CN Electronic cigarette 15 mg
Device: Nicorette Inhalator 15 mg — Inhalation
  Arms: Nicorette Inhalator 15 mg
Other: Cigarette — Inhalation
  Arms: Cigarette

SUMMARY:
The purpose of this study is to assess the amount of nicotine that is absorbed into the blood stream following the use of a new Electronic Cigarette device called the CN electronic cigarette. The amount of nicotine delivered via the CN electronic cigarette will be compared to the amount of nicotine delivered from smoking a regular cigarette and from using the Nicorette® Inhalator.

Electronic cigarettes aim to mimic the experience of cigarette smoking, by delivering nicotine rapidly. Unlike cigarettes however, they do not contain all of the many harmful combustion products contained in tobacco smoke.

Electronic cigarettes are readily available in many markets, and may contain significant quantities of nicotine. However, they are not regulated as medicines, and their manufacturers can make no medicinal claims about them.

Such products are unregulated, having not been subjected to regulatory review by either the Medicines and Healthcare Products Regulatory Agency (MHRA) or any Notified Body.

It is the intention of CN Creative (makers of the CN electronic cigarette) to submit an application to the MHRA for the CN Electronic Cigarette, in order to make a high quality, regulated product available. Males aged 18-65, who smoke and who have no intention of stopping smoking during the trial are eligible to take part in this study. The study consist of a screening visit, a treatment period with 5 overnight stays with nicotine treatment on days 1, 2, 3 and 4 with a post study visit on day 5.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed written informed consent.
* Males aged 18-65 years.
* Subject with a Body Mass Index (BMI) of 18-30 Body Mass Index = Body weight (kg) / [Height (m)]2.
* Regular moderate cigarette smokers (approximately 10 to 20 cigarettes per day for at least 5 years) who are not intending to make a quit attempt during the study.
* No obvious symptoms of ill health as determined during the pre-study medical examination (to be performed within 4 weeks of the first dose).
* Subject with no clinically significant abnormalities in 12-lead electrocardiogram (ECG), including normal resting ECG with QTcB interval of less than 440 ms determined within 4 weeks of the first dose.
* No clinically significant abnormalities in blood pressure values (the differences between supine and standing BP are less than 20 mmHg) with no symptomatic evidence of postural hypotension.
* Subject with no clinically significant abnormal serum biochemistry, haematology and urine examination values within 4 weeks of the first dose.
* Subject with a negative urinary drugs of abuse screen (excluding nicotine), determined within 4 weeks of the first dose (N.B. a positive alcohol result may be repeated at the discretion of the Investigator).
* Subject with negative HIV and Hepatitis B and C results.

To be re-confirmed at Day 0:

* Subject continues to meet all screening inclusion criteria.
* Subject with a negative urinary drugs of abuse screen (including alcohol) prior to dosing

Exclusion Criteria:

* To be confirmed at Screening Visit:
* Evidence of renal, hepatic, central nervous system, respiratory (including COPD), cardiovascular or metabolic dysfunction.
* Known allergy to any ingredients of the study medication.
* A history of or current drug or alcohol abuse.
* Inability to communicate well with the Investigator/study staff (i.e., language problem, poor mental development or impaired cerebral function).
* Participation in a New Chemical Entity clinical study within the previous 4 months or a marketed drug clinical study within the previous 3 months (N.B. washout period between trials defined as the period of time elapsed between the last dose of the previous study and the first dose of the next study..
* Donation of 450ml or more blood within the previous 3 months.
* Any other clinically significant medical history, in theInvestigator's opinion, including conditions which might affect drug absorption, metabolism or excretion.
* Unlikely to comply with trial visit schedule or with trial medication dosing requirements.
* Severe intercurrent illness which, in the opinion of the Investigator, may put the subject at risk when participating in the trial or may influence the results of the trial or affect the subjects' ability to take part in the trial.
* Excessive intake of alcohol, defined as a regular maximum weekly intake of greater than 28 units for men (1 unit equals half a pint of beer, 1 small glass of wine or 1 x 25 mL measure of spirits) within the last 6 months.
* Treatment with smoking cessation medications (bupropion, Champix, any NRT) within 8 weeks of the planned first nicotine dosing occasion.
* Treatment with prescription medications within 21 days or over-the-counter medication within 72 hours of the planned first nicotine dosing occasion.
* Clinical judgement by the Investigator that the subject should not participate in the study for any other reason.

To be re- confirmed at Day 0:

* Development of any exclusion criteria since screening
* Receipt of any medication since screening visit that may have an impact on the safety and objectives of the study (at the Investigator's discretion).

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-08; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Cmax: The peak serum concentration of nicotine. | 0 to 20h, PK parameters calculated after 4th Administration
  PK samples taken after 4th administration immediately after dosing and 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 30, 60 minutes, and 2, 4, 6, 8, 12 and 20 hours afterwards. The pre-dose blood sample drawn on days 2, 3 and 4 will also serve as the 20 hour sample

SECONDARY OUTCOMES:
AUC0-t | 0 to 20h, PK parameters calculated after 4th Administration
Tmax | 0 to 20h, PK parameters calculated after 4th Administration
t½ | 0 to 20h
Cmin | 0 to 20h, PK parameters calculated after 4th Administration

CONTACTS AND LOCATIONS:
Overall Officials: Girish Sharma, MBBS, Principal Investigator — Simbec Research

IPD SHARING:
Plan to Share IPD: Yes
Yes, data has been shared on EudRACT in the form of a poster presentation. Sharma G, Lawson D, Edwards C et al. A Novel Electronic Cigarette with Advanced Vaporization Technology: Nicotine Pharmacokinetics (PK), Safety and Tolerability. Poster presentation at 21st Annual Meeting of the Society of Research on Nicotine and Tobacco (SRNT); Philadelphia, USA; February 25 - 28 2015